CLINICAL TRIAL: NCT06030024
Title: An Open-lable Investigation of the Effect of rTMS on Attention in an Adult Sample Suffering From ADD
Brief Title: Efficacy of Repetitive Transcranial Magnetic Stimulation in Adult Attention Deficit Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tehran (Other)
Responsible Party: Principal Investigator, reza kazemi, Assistant professor, University of Tehran
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Attention
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Attention Deficit Disorder; ADHD
Keywords: rTMS; ADHD; ADD; fMRI
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active rTMS (Experimental): Participants in this one and only arm in the current study received active repetitive transcranial magnetic stimulation.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation — Magnetic pulses delivered to the Fz area of the brain in a low frequency (1 Hz) manner.

SUMMARY:
The purpose of the current open-lable study was to use low-frequency repetitive transcranial magnetic stimulation (rTMS) to improve the attention deficits in a sample of adult patients suffering from attention deficit disorder. Participants received 10 sessions of rTMS over Fz (located using the EEG 10-20 international system) and underwent assessments of their attentional capacity using the gradCPT task in an fMRI scanner, before and after the intervention. Other behavioral assessments of their attention symptoms have also been conducted.

ELIGIBILITY:
Inclusion Criteria:

* Normal intelligence level (>90)
* Diagnosis of ADD by a psychiatrist using the ADHD-RS-IV with Adult Prompts

Exclusion Criteria:

* Scores of 21 or more on BDI and/or BAI
* History of head trauma
* History of a major psychological or neurological condition
* Presence of metal in the head
* History of seizures
* Serious cardiovascular disease
* Use of medications with an impact on cognitive functions during the treatment window (patients with a constant and stable dose were included)
* Recent use of alcohol or substance abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Change in performance | Up to 10 days, i.e., before and after the completion of the 10 sessions of rTMS
  Shortened version (4 min) of the continuous go/no-go task: gradual-onset continuous performance task (gradCPT)

SECONDARY OUTCOMES:
Change in self-report attention scores | Baseline, after 5 days of stimulation, after 10 days of stimulation; Range= 0-6; Higher scores represent worse outcome
  The 6-item ASRS-V1.1 Adult ADHD Self-Report
Change in investigator-rated attention scores | Baseline, after 5 days of stimulation, after 10 days of stimulation; Range:0 - 54; Higher scores represent worse outcome
  Investigator-Rated Attention-Deficit Hyperactivity Disorder (ADHD) Rating Scale-IV (I-ADHD RS-IV) with adult prompts

CONTACTS AND LOCATIONS:
Overall Officials: Reza Rostami, M.D, Study Director — University of Tehran; Fatemeh Soltani, MSc, Principal Investigator — University of Tehran
Locations (1):
- National Brain Mapping Lab, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No